CLINICAL TRIAL: NCT06282913
Title: The Effect of Mindfulness Meditation Practice on Compassion Fatigue, Burnout, and Psychological Well-Being of Health Professionals Working in Oncology Units: Randomized Controlled Study
Brief Title: The Effect of Mindfulness Meditation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gulhane Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Buğse Yüceer, Phd Student, Gulhane Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ---Oncology-Nursing-2024---
Record Dates: First submitted 2024-01-09; First posted 2024-02-28 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Burnout; Compassion Fatigue; Psychological Well-Being
Keywords: Mindfulness meditation; compassion fatigue; burnout; psychological well-being; oncology units; health professionals
MeSH Terms: conditions — Burnout, Psychological; Compassion Fatigue; Psychological Well-Being | interventions — Mindfulness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mindfulness Meditation Group (Experimental): During the first meeting, before the planned training, data will be collected face to face using the personal information form, Compassion Fatigue Brief Scale, Maslach Burnout Scale, Psychological Well-Being Scale. Physicians and nurses in the intervention group were given group counseling sessions by the researcher, in groups of 10-15 people, for 20 minutes once a week for 8 weeks. An online meditation practice will be provided for a long time. At the end of the mindfulness meditation application (in the 8th week) and four weeks after the end of the application (in the 12th week) for follow-up purposes, data will be collected through an online survey for physicians and nurses using Compassion Fatigue Brief Scale, Maslach Burnout Scale, Psychological Well-Being Scale.
  Interventions: Behavioral: Mindfulness Meditation
- Control Group (No Intervention): During the first meeting, data will be collected face to face using the personal information form, MY-KÖ, MTÖ and PİÖÖ. In the 8th and 12th weeks of the research, the data will be re-administered to the physicians and nurses in the control group via an online survey using Compassion Fatigue Brief Scale, Maslach Burnout Scale, Psychological Well-Being Scale. After the implementation process of the research is completed, mindfulness meditation application will be applied online once to the physicians and nurses in the control group.

INTERVENTIONS:
Behavioral: Mindfulness Meditation — Mindfulness Meditation application will be implemented online by the researcher in 20-minute group sessions once a week for 8 weeks. Participants will be asked to provide a quiet, ventilated, dimly lit environment for the practice. The researcher will start the application when the participants take their places as they feel comfortable. In the first stage, the researcher will teach physicians and nurses to take deep diaphragmatic breaths through the nose and out through the mouth.
  Arms: Mindfulness Meditation Group

SUMMARY:
Cancer is a disease that causes the most deaths worldwide and is challenging for patients and caregivers both physically and psychosocially. Physicians and nurses working in oncology clinics perform a demanding profession providing compassionate care and treatment to patients struggling with life-threatening diseases. The emotional cost of caring for patients diagnosed with cancer can lead to compassion fatigue, burnout, and decreased psychological well-being among healthcare professionals. For this reason, this research is planned as a randomized controlled study to examine the effect of Mindfulness meditation practice on compassion fatigue, burnout, and psychological well-being in physicians and nurses working in oncology units.

ELIGIBILITY:
Inclusion Criteria:

* Actively working in oncology clinics
* At least 1 year of working experience in an oncology clinic
* Not having a physical/mental/psychological disorder that would prevent participation in the research.
* Oncology nurses with a high school, undergraduate, associate or graduate degree in nursing
* Physicians and nurses who volunteer to participate in the research will be included in the research sample.

Exclusion Criteria:

* Physicians and nurses who have been diagnosed with a psychological disease in the last two years and are continuing their medical treatment • Physicians and nurses who did not agree to participate in the research

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
compassion fatigue | up to 8 weeks
  At the end of the mindfulness meditation practice in oncology physicians and nurses the Compassion Fatigue Brief Scale will be used to measure the changes in compassion fatigue. As the scores obtained from the compassion fatigue brief scale increase, the perceived level of compassion fatigue in individuals increases. The lowest score from the scale is 13 and the highest score is 130.
burnout | up to 8 weeks
  At the end of the mindfulness meditation practice in oncology physicians and nurses the Maslach Burnout Scale will be used to measure the changes in the level of burnout. Increasing Maslach Burnout Scale "Depersonalization" and "Emotional exhaustion" subscale scores indicate that burnout increases, while increasing the "personal success" subscale score indicates that burnout decreases.
psychological well-being | up to 8 weeks
  At the end of the mindfulness meditation practice in oncology physicians and nurses and the Psychological Well-Being Scale will be used to evaluate the changes in the level of psychological well-being. A high score on the psychological well-being scale indicates that the person is at a positive level psychologically. The highest score from the scale is 56, while the minimum score is 8.

SECONDARY OUTCOMES:
compassion fatigue | up to 12 weeks
  Four weeks after the end of the mindfulness meditation practice in oncology physicians and nurses the Compassion Fatigue Brief Scale will be used to measure the changes in compassion fatigue. As the scores obtained from the compassion fatigue brief scale increase, the perceived level of compassion fatigue in individuals increases. The lowest score from the scale is 13 and the highest score is 130.
burnout | up to 12 weeks
  Four weeks after the end of the mindfulness meditation practice in oncology physicians and nurses the Maslach Burnout Scale will be used to measure the changes in the level of burnout. Increasing Maslach Burnout Scale "Depersonalization" and "Emotional exhaustion" subscale scores indicate that burnout increases, while increasing the "personal success" subscale score indicates that burnout decreases.
psychological well-being | up to 12 weeks
  Four weeks after the end of the mindfulness meditation practice in oncology physicians and nurses and the Psychological Well-Being Scale will be used to evaluate the changes in the level of psychological well-being. A high score on the psychological well-being scale indicates that the person is at a positive level psychologically. The highest score from the scale is 56, while the minimum score is 8.

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Abdurrahman Yurtaslan Oncology Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No